CLINICAL TRIAL: NCT01203852
Title: Pharmacogenomic Evaluation of Antihypertensive Responses 2
Acronym: PEAR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201700661-N; U01GM074492-06 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: hypertension; antihypertensive drug; pharmacogenetics; genetics; blood pressure; glucose
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metoprolol + Chlorthalidone (Experimental): Study participants in this group had their current hypertension treatment withdrawn, baseline labs drawn and hypertension documented. Participants were initiated on metoprolol tartrate 50 mg twice daily for two weeks, followed by dose titration to 100 mg twice daily for six additional weeks if blood pressure (BP) > 120/70 mmHg. BP measures were again recorded. Participants entered a washout where metoprolol was titrated, then discontinued, and the patient's hypertension was re-established. After another set of identical baseline labs, study participants were initiated on chlorthalidone 25 mg four days per week (Monday, Wednesday, Thursday, Saturday) 15 mg daily for two weeks, followed by 25 mg daily for an additional six weeks.
  Interventions: Drug: Metoprolol; Drug: Chlorthalidone

INTERVENTIONS:
Drug: Metoprolol — Metoprolol 50 mg twice daily titrated to 100 mg twice daily
  Note: due to discontinuation of the manufacture of chlorthalidone 15 mg, effective Jan 1, 2013; the starting dose of chlorthalidone will be 25 mg 4 times per week (Mon, Wed, Thur, Sat) with subsequent titration to 25 mg daily.
  Other Names: Lopressor; Toprol XL
Drug: Chlorthalidone — Chlorthalidone 25 mg 4 times per week titrated to 25 mg daily
  Other Names: Thalitone

SUMMARY:
There are many medications available for the treatment of high blood pressure (hypertension), but finding the right one for a specific patient can be challenging. In fact, it is estimated that less than 50% of people with hypertension have their blood pressure under control. The hypothesis is that genetic differences between individuals influence their response to antihypertensive medications. This study is aimed at determining the genetic factors that may influence a person's response to either a beta-blocker or a thiazide diuretic. The hope is that through this research, the investigators may someday be able to use an individual's genetic information to guide the selection of their blood pressure medicine, leading to better control of blood pressure, and less need for the current trial and error process.

DETAILED DESCRIPTION:
The proposed work should help move toward the long-term goal of selection of antihypertensive drug therapy based on a patient's genetic make-up. Hypertension (HTN) is the most common chronic disease for which drugs are prescribed, and the most prevalent risk factor for heart attack, stroke, renal failure and heart failure. Responses to antihypertensive drug therapy exhibit considerable interpatient variability, contributing to poor rates of HTN control (currently about 40-50% in the US), and frequent nonadherence and dropout from therapy. We propose to identify genetic predictors of the antihypertensive and adverse metabolic responses to two preferred and pharmacodynamically contrasting drugs, a beta-blocker (metoprolol) and a thiazide diuretic (chlorthalidone) in a sequential monotherapy design in 400 hypertensive individuals. Data collected will include home and clinic blood pressure, blood samples for testing for adverse metabolic effects and other biomarkers, RNA, and DNA and urine sample. We will conduct genome-wide association single nucleotide polymorphism (SNP) genotyping and data from the study will be used for replication of findings from the previous PEAR trial, along with new discoveries. The primary aims are to define the genetic determinants of the antihypertensive response and adverse metabolic responses (e.g. changes in glucose, triglycerides and uric acid). The proposed research is significant because genetically-targeted antihypertensive therapy could lead to dramatically higher response rates and fewer adverse effects than the usual trial-and-error approach. This would likely lead to higher rates of HTN control, less need for polypharmacy, reduced health care costs, and improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* An average seated home diastolic blood pressure (DBP) > 85 mmHg and < 110 mmHg and home systolic blood pressure (SBP) < 180 mmHg.
* Subjects must also have an average seated (> 5 minutes) clinic DBP between 90 mmHg and 110 mmHg and SBP < 180 mmHg

Exclusion Criteria:

* Secondary forms of hypertension (HTN) (including sleep apnea)
* Isolated systolic HTN
* Other diseases requiring treatment with BP lowering medications
* Heart rate < 55 beats/min (for metoprolol only)
* Known cardiovascular disease (including history of angina pectoris, heart failure, presence of a cardiac pacemaker, history of myocardial infarction or revascularization procedure, or cerebrovascular disease, including stroke and TIA)
* Diabetes mellitus (Type 1 or 2)
* Renal insufficiency (serum creatinine > 1.5 in men or 1.4 in women)
* Primary renal disease
* Pregnancy or lactation
* Liver enzymes > 2.5 upper limits of normal
* Current treatment with NSAIDS, cyclooxygenase-2 (COX2) inhibitors, oral contraceptives or estrogen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, PharmD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Mayo Clinic, Division of Hypertension, Rochester, Minnesota

REFERENCES:
- [Background] Hamadeh IS, Langaee TY, Dwivedi R, Garcia S, Burkley BM, Skaar TC, Chapman AB, Gums JG, Turner ST, Gong Y, Cooper-DeHoff RM, Johnson JA. Impact of CYP2D6 polymorphisms on clinical efficacy and tolerability of metoprolol tartrate. Clin Pharmacol Ther. 2014 Aug;96(2):175-81. doi: 10.1038/clpt.2014.62. Epub 2014 Mar 17. PMID 24637943
- [Derived] Mehanna M, McDonough CW, Smith SM, Gong Y, Gums JG, Chapman AB, Johnson JA, Cooper-DeHoff RM. Integrated metabolomics analysis reveals mechanistic insights into variability in blood pressure response to thiazide diuretics and beta blockers. Clin Transl Sci. 2024 May;17(5):e13816. doi: 10.1111/cts.13816. PMID 38747311
- [Derived] Chekka LMS, Tantawy M, Langaee T, Wang D, Renne R, Chapman AB, Gums JG, Boerwinkle E, Cooper-DeHoff RM, Johnson JA. Circulating microRNA Biomarkers of Thiazide Response in Hypertension. J Am Heart Assoc. 2024 Feb 20;13(4):e032433. doi: 10.1161/JAHA.123.032433. Epub 2024 Feb 14. PMID 38353215
- [Derived] Mehanna M, Wang Z, Gong Y, McDonough CW, Beitelshees AL, Gums JG, Chapman AB, Schwartz GL, Bailey KR, Johnson JA, Turner ST, Cooper-DeHoff RM. Plasma Renin Activity Is a Predictive Biomarker of Blood Pressure Response in European but not in African Americans With Uncomplicated Hypertension. Am J Hypertens. 2019 Jun 11;32(7):668-675. doi: 10.1093/ajh/hpz022. PMID 30753254
- [Derived] Sa ACC, Webb A, Gong Y, McDonough CW, Shahin MH, Datta S, Langaee TY, Turner ST, Beitelshees AL, Chapman AB, Boerwinkle E, Gums JG, Scherer SE, Cooper-DeHoff RM, Sadee W, Johnson JA. Blood pressure signature genes and blood pressure response to thiazide diuretics: results from the PEAR and PEAR-2 studies. BMC Med Genomics. 2018 Jun 20;11(1):55. doi: 10.1186/s12920-018-0370-x. PMID 29925376
- [Derived] Singh S, McDonough CW, Gong Y, Alghamdi WA, Arwood MJ, Bargal SA, Dumeny L, Li WY, Mehanna M, Stockard B, Yang G, de Oliveira FA, Fredette NC, Shahin MH, Bailey KR, Beitelshees AL, Boerwinkle E, Chapman AB, Gums JG, Turner ST, Cooper-DeHoff RM, Johnson JA. Genome Wide Association Study Identifies the HMGCS2 Locus to be Associated With Chlorthalidone Induced Glucose Increase in Hypertensive Patients. J Am Heart Assoc. 2018 Mar 9;7(6):e007339. doi: 10.1161/JAHA.117.007339. PMID 29523524
- [Derived] Shahin MH, Sa AC, Webb A, Gong Y, Langaee T, McDonough CW, Riva A, Beitleshees AL, Chapman AB, Gums JG, Turner ST, Boerwinkle E, Scherer SE, Sadee W, Cooper-DeHoff RM, Johnson JA. Genome-Wide Prioritization and Transcriptomics Reveal Novel Signatures Associated With Thiazide Diuretics Blood Pressure Response. Circ Cardiovasc Genet. 2017 Jan;10(1):e001404. doi: 10.1161/CIRCGENETICS.116.001404. PMID 28115488
- See also: PEAR study website — http://www.pear.cop.ufl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was recruited on 8/10/10 and the final patient was recruited on 9/30/2013. Subjects were recruited from family medicine clinics and were identified through providers daily schedules, medical records, and encounter forms.
Pre-assignment Details: Healthy volunteers with mild to moderate primary hypertension between the ages of 18-70 were eligible for the study. Subjects were washed-out from their hypertension medication prior to beginning study protocol. Participants with elevated systolic blood pressure greater than 180 mmHg after wash-out were excluded from the study.
Groups:
- Metoprolol + Chlorthalidone: This group was assigned the following:
  (Metoprolol 8 weeks): Metoprolol tartrate 50 mg twice daily for two weeks. After two weeks subjects will be seen in clinic and will have the dose doubled to 100 mg twice daily if either their home blood pressure (HBP) average or office blood pressure (OBP) is > 120/70 mmHg. They will continue on this dose for an additional 6 weeks.
  (Washout 2 weeks): Then will washout from all study medication.
  (Chlorthalidone 8 weeks): participants will initiate chlorthalidone 25 mg four times per week (Monday, Wednesday, Thursday, Saturday) for two weeks, then 25 mg daily of chlorthalidone for 6 weeks.
Period: Metoprolol 8 Weeks
Arm/Group | Metoprolol + Chlorthalidone
Started | 839 (This is the total number of subjects for both groups.)
Completed | 369
Not Completed | 470
Not completed — Physician Decision | 470
Period: Washout 2 Weeks
Arm/Group | Metoprolol + Chlorthalidone
Started | 328 (Some study subjects did not proceed to the washout phase after the first intervention.)
Completed | 282
Not Completed | 46
Not completed — Physician Decision | 46
Period: Chlorthalidone 8 Weeks
Arm/Group | Metoprolol + Chlorthalidone
Started | 328 (Subjects were allowed to enter the study at Chlorthalidone without completing Metoprolol.)
Continued From Metoprolol | 282
Completed | 328
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Approximately 1000 males or females with mild to moderate primary HTN, of any race or ethnicity, between the ages of 18 and 65 will be enrolled into the PEAR2 protocol. Prospective study participants will be those with newly diagnosed HTN, untreated HTN or known HTN currently treated with antihypertensive drugs.
Groups:
- Metoprolol + Chlorthalidone: This group was assigned to the following: Metoprolol tartrate 50 mg twice daily for two weeks. After two weeks subjects will be seen in clinic and will have the dose doubled to 100 mg twice daily if either their HBP average or OBP is > 120/70 mmHg. They will continue on this dose for an additional 6 weeks. Then will washout from all study medication. After washout, participants will initiate chlorthalidone 25 mg four times per week (Monday, Wednesday, Thursday, Saturday) for two weeks, then 25 mg daily of chlorthalidone for 6 weeks.
  Metoprolol: Metoprolol 50 mg twice daily titrated to 100 mg twice daily
  Chlorthalidone: Chlorthalidone 25 mg 4 times per week titrated to 25 mg daily
  Note: due to discontinuation of the manufacture of chlorthalidone 15 mg, effective Jan 1, 2013; the starting dose of chlorthalidone will be 25 mg 4 times per week (Mon, Wed, Thur, Sat) with subsequent titration to 25 mg daily.
Arm/Group | Metoprolol + Chlorthalidone
Number analyzed (Participants) | 839
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 839
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429
  Male | 410
Region of Enrollment [Number; unit: participants]
  United States | 839

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure From Baseline to Treatment
Description: Response to blood pressure medication will be assessed by measuring blood pressure before and after treatment
Time Frame: after 6-8 weeks of treatment
Population: All patients with antihypertensive response data. 282 patients completed all 3 study periods. 369 patients completed only period 1. 328 patients completed only period 3.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Metoprolol + Chlorthalidone: Study participants had their current hypertension treatment withdrawn, baseline labs drawn and hypertension documented. Participants were initiated on metoprolol tartrate 50 mg twice daily for two weeks, followed by dose titration to 100 mg twice daily for six additional weeks if blood pressure (BP) > 120/70 mmHg. BP measures were again recorded. Participants entered a washout where metoprolol was titrated, then discontinued, and the patient's hypertension was re-established. After another set of identical baseline labs, study participants were initiated on chlorthalidone 25 mg four days per week (Monday, Wednesday, Thursday, Saturday) 15 mg daily for two weeks, followed by 25 mg daily for an additional six weeks.
- Metorprolol Only: Study participants had their current hypertension treatment withdrawn, baseline labs drawn and hypertension documented. Participants were initiated on metoprolol tartrate 50 mg twice daily for two weeks, followed by dose titration to 100 mg twice daily for six additional weeks if blood pressure (BP) > 120/70 mmHg. BP measures were again recorded.
- Chlorthalidone Only: Study participants were initiated on chlorthalidone 25 mg four days per week (Monday, Wednesday, Thursday, Saturday) 15 mg daily for two weeks, followed by 25 mg daily for an additional six weeks.
Arm/Group | Metoprolol + Chlorthalidone | Metorprolol Only | Chlorthalidone Only
Number analyzed (Participants) | 282 | 369 | 328
mmHg
  diastolic blood pressure response | -7.56 (6.39) | -7.97 (6.48) | -7.68 (5.84)
  systolic blood pressure response | -11.70 (9.51) | -7.45 (9.85) | -13.65 (9.55)
Statistical Analysis 1: Comparison: Metoprolol + Chlorthalidone; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value for one sided t-test of mean change in blood pressure before and after treatment with metoprolol and chlorthalidone were <0.0001

2. Secondary Outcome: Adverse Metabolic Effects
Description: Change in glucose after treatment with study medication
Time Frame: after 6-8 weeks treatment
Population: All patients with change in glucose data
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Adverse Metabolic Effects: Change in glucose after treatment with study medications
Arm/Group | Adverse Metabolic Effects
Number analyzed (Participants) | 365
mg/dL
  glucose response to metoprolol (n=365) | 1.02 (9.83)
  glucose response to chlorthalidone (n=318) | 5.12 (10.6)
Statistical Analysis 1: Comparison: Adverse Metabolic Effects; Mean glucose change after treatment with chlorthalidone; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value for one sided t-test for mean glucose change before and after treatment with chlorthalidone was <0.0001
Statistical Analysis 2: Comparison: Adverse Metabolic Effects; Mean glucose change after treatment with metoprolol; Test type: Superiority or Other; p = 0.049, t-test, 1 sided — P-value for one sided t-test for mean glucose change before and after treatment with metoprolol was 0.049

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during subject participation in the study. Participation lasted between 3 and 4 months.
Description: Adverse events were not recorded according to intervention.
Groups:
- All Study Participants: Study participants had their current hypertension treatment withdrawn, baseline labs drawn and hypertension documented. Participants were initiated on metoprolol tartrate 50 mg twice daily for two weeks, followed by dose titration to 100 mg twice daily for six additional weeks if blood pressure (BP) > 120/70 mmHg. BP measures were again recorded. Participants entered a washout where metoprolol was titrated, then discontinued, and the patient's hypertension was re-established. The subjects were initiated on chlorthalidone 25 mg four days per week (Monday, Wednesday, Thursday, Saturday) 15 mg daily for two weeks, followed by 25 mg daily for an additional six weeks.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 3/839
Other Adverse Events (participants affected / at risk) | 114/839
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=839)
Headache (Vascular disorders) | 2 (2)
Heart Attack (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=839)
Bradycardia (Cardiac disorders) | 2 (2)
Chest Pain (Cardiac disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Ear and labyrinth disorders) | 10 (11)
Dyspnea (Nervous system disorders) | 1 (1)
Headache (Vascular disorders) | 29 (32)
Nausea (Gastrointestinal disorders) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Fatigue (General disorders) | 15 (16)
Other (General disorders) | 41 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No